CLINICAL TRIAL: NCT04703790
Title: Acceptability Across Two Time Periods of a SARS-CoV-2 Vaccine Among a Representative Sample of Adults Within the United States
Brief Title: Acceptability of a COVID-19 Vaccine Among US Adults Over Two Time Periods
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Susan Rosenthal, PhD, ABPP, Professor of Medical Psychology (in Pediatrics and Psychiatry), Columbia University
Other Study IDs: AAAT5154
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Vaccine Acceptability
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults from the United States: Adult participants 18 years of age or older who are panelists recruited and maintained by Ipsos (KnoweledgePanel). All participants live within the United States.

SUMMARY:
The overall purpose of this study is to address the factors associated with an individual's personal willingness to get the vaccine and attitudes about potential public policy approaches to implementation of a Coronavirus Disease 2019 (COVID-19) vaccine. Additionally, to evaluate how these attitudes change over time. The 1200 participants will be recruited by Ipsos (Ipsos KnowledgePanel®) from their nationally representative panel to participate in a survey at Time 1 and 1 year later. The information collected will include demographics, health status, household composition, experiences with COVID-19, attitudes about vaccines in general, COVID-19 vaccine specific attitudes, willingness to get a COVID-19 vaccine acceptability, and attitudes regarding COVID-19 vaccine mandates. The investigators anticipate that those who live in urban areas and who are older, have greater knowledge of COVID-19, who have known someone who was hospitalized for COVID-19, and have generally positive attitudes about vaccines will be more willing to get a vaccine. The primary reasons for willingness will be personal safety and desire to return to normal activities. The investigators also anticipate that those who vary on socio-demographics (e.g., live in urban areas, have more liberal political views), have greater knowledge of COVID-19, who have known someone who was hospitalized for COVID- 19, and have generally positive attitudes about vaccines will be more supportive of mandatory vaccination strategies. The investigators anticipate that attitudes will change over time in response to the current status of the pandemic and of available data about the vaccine's efficacy and safety.

DETAILED DESCRIPTION:
The overall objective is to address attitudes about potential public policy approaches to implementation of a Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) vaccine and the factors associated with an individual's personal willingness to get the vaccine once available, and to assess how these attitudes change over time.

First specific aim:

1a. To describe participants' perceptions of public health strategies including mandatory vaccination requirements (e.g., travel, school attendance, work place requirements (e.g., schools, health care facilities, offices), working in a health care facility, health care providers, living in residential facilities) and targeted age groups (e.g., children, adolescents, adults, elderly).

1. b. To determine how attitudes about strategies are related to socio-demographic characteristics (e.g., age, education, race/ethnicity, political views and political party affiliation, household structure), knowledge of SARS-CoV-2, personal experience with the infection, and other vaccine attitudes.

   Example hypothesis: Those who vary on socio-demographics (e.g., live in urban areas, have more liberal political views), have greater knowledge of SARS-CoV-2, who have known someone who was hospitalized for SARS-CoV-2, and have generally positive attitudes about vaccines will be more supportive of mandatory vaccination strategies.

   Second specific aim:
2. a. To determine the relationship of socio-demographic characteristics (e.g., age, education, race/ethnicity, political views and political party affiliation, household structure), knowledge of SARS-CoV-2, personal experience with the infection, and other vaccine attitudes with willingness to get the vaccine.

2b. To evaluate the primary reasons driving vaccine acceptance including safety issues (personal, family, or global), desire to return to normal activities (e.g., school, work, or social events), and desire to no longer need to wear a mask.

Example hypotheses: Those who vary on socio-demographic characteristics (e.g., live in urban areas, who are older), have greater knowledge of SARS-CoV-2, who have known someone who was hospitalized for SARS-CoV-2, and have generally positive attitudes about vaccines will be more willing to get a vaccine. The primary reasons for willingness will be personal safety and desire to return to normal activities.

Third specific aim: This specific aim focuses on how the findings from aim 1 and aim 2 change over time.

3a. To evaluate how national level perceptions of public health strategies (aim 1) and an individual's personal willingness to get the vaccine (aim 2) change over time.

Given the unknown trajectory, there are several possible scenarios. For example, if nationally there is a decrease in new infections with lifting of the restrictions then the investigators hypothesize that there will be an overall decrease in support for mandatory strategies and in willingness to accept the vaccine. Alternatively, if new infections are rising and restrictions are in place, then there will be an overall increase in acceptability. The investigators are also prepared to adapt our surveys should one or more vaccines become licensed and available prior to the time 1 or time 2 survey.

3b. The investigators will explore whether changes in perceptions of public health strategies (aim 1) and an individual's personal willingness to get the vaccine (aim 2) vary based on relevant socio-demographic characteristics (e.g., region of the country, political views and political party affiliation, household structure, race/ethnicity) and, when appropriate, changes within those characteristics (e.g., when rates of infections are changing differentially across regions). The investigators also will explore whether changes in perceptions of public health strategies (aim 1) and an individual's personal willingness to get the vaccine (aim 2) vary based on perceptions of societal events. For example, the investigators will evaluate if changes in vaccine attitudes are associated with regional differences in whether cases are increasing or decreasing; changes in household structure (e.g., the presence of elders in the home); or perceptions of media reports.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Able to read English and Spanish
* Panelists with Ipsos (KnowledgePanel)

Exclusion Criteria:

* 17 years of age and younger
* Not able to read English or Spanish
* Not a member of Ipsos (KnowledgePanel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years of age and older, who live in the US and who have been recruited to be members of Ipsos (KnowledgePanel) survey research panel.
Sampling Method: Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Vaccination or intention to get vaccinated for COVID-19 | Baseline, 1 year
  Participants vaccination status or intent to get vaccinated for COVID-19 will be measured via survey items.

SECONDARY OUTCOMES:
Attitudes toward mandates for COVID-19 vaccines | Baseline, 1 year
  Participants self report of attitudes on survey

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Rosenthal, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No